CLINICAL TRIAL: NCT01371643
Title: Does Surgical Debulking Of Pituitary Adenomas Improve Responsiveness To Octreotide LAR In The Treatment Of Acromegaly: An Investigator-Initiated Study
Brief Title: Surgical Debulking of Pituitary Adenomas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R11104
Record Dates: First submitted 2011-06-09; First posted 2011-06-13 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Pituitary Adenoma
MeSH Terms: conditions — Pituitary Neoplasms

ARMS (2):
- Medical treatment by Octreotide LAR (Active Comparator): Medical therapy with Octreotide LAR 30 mg/month for 3 months preceding surgery
  Interventions: Drug: Octreotide LAR
- Surgical debulking followed by Octreotide LAR (Active Comparator): Surgical debulking of pituitary tumor followed by Octreotide LAR if not surgically cured
  Interventions: Drug: Octreotide LAR; Procedure: transsphenoidal surgery

INTERVENTIONS:
Drug: Octreotide LAR
Procedure: transsphenoidal surgery
  Arms: Surgical debulking followed by Octreotide LAR

SUMMARY:
This is a randomized, multicenter trial with stratification done by a single radiologist at the coordinating center (NYU), and patients with comparable disease will be randomized to Sandostatin LAR treatment administered 1 time per month by IM injection for 3 months before (Arm A) or, for non-cured patients, after (Arm B) surgery. All patients will undergo transsphenoidal hypophysectomy. The impact of surgical debulking on responsiveness to Sandostatin LAR will be evaluated.The primary objective of this trial will be to determine whether surgery (debulking of pituitary adenomas) improves the response of patients with acromegaly to treatment with Octreotide LAR, when compared to Octreotide LAR therapy alone.

DETAILED DESCRIPTION:
The current goal of treatment for people with acromegaly is normalization of both growth hormone (GH) and insulin-like-growth-factor-1 (IGF-1) levels. Normalization of GH and IGF-1 levels attenuates the morbidity (hypertension, cardiovascular disease, sleep apnea, increased cancer risk, arthritis) and increased mortality associated with persistent GH and IGF-1 elevation. The optimal approach to achieving these goals in patients with pituitary macroadenomas remains controversial. Available treatment modalities include transsphenoidal hypophysectomy, medical therapy (somatostatin analogues and/or dopaminergic agonists), radiotherapy, or a combination or these interventions. No randomized trials have been conducted to investigate whether surgical debulking of pituitary macroadenomas enhances the efficacy of medical therapy. This study is designed to rigorously investigate whether surgical debulking increases the efficacy of a long-acting depot somatostatin preparation, Sandostatin LAR, so that evidence-based optimal care may be offered to patients with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Carry a diagnosis of de novo acromegaly with an elevated age and sex matched IGF-I and GH >1ng/ml at all time points during OGTT
* Have a pituitary macroadenoma
* Have clinical changes consistent with acromegaly
* Have a single random serum hGH of 12.5 ng/ml or greater
* Both the endocrinologist and surgeon must agree that the patient's health would not be compromised by a three-month period during which time Octreotide LAR is administered.
* Patients currently on dopamine agonist who agree to discontinue medication (2-6 week washout required)

Exclusion Criteria:

* Pregnant or breastfeeding
* Documented loss of vision due to pituitary tumor
* Prior treatment for acromegaly other than dopamine agonists
* Inability to complete the protocol
* Intolerance to octreotide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2004-04; Primary Completion 2010-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Kleinberg, MD, Principal Investigator — NYU School of Medicine
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Treatment by Octreotide LAR: Medical therapy with Octreotide LAR 30 mg/month for 3 months preceding surgery
  Octreotide LAR
- Surgical Debulking Followed by Octreotide LAR: Surgical debulking of pituitary tumor followed by Octreotide LAR if not surgically cured
  Octreotide LAR
  transsphenoidal surgery
Period: Overall Study
Arm/Group | Medical Treatment by Octreotide LAR | Surgical Debulking Followed by Octreotide LAR
Started | 15 | 26
Completed | 12 | 26
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Treatment by Octreotide LAR | Surgical Debulking Followed by Octreotide LAR | Total
Number analyzed (Participants) | 15 | 26 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 25 | 39
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 10 | 14 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaskan | 0 | 0 | 0
  Asian or Pacific Islander | 1 | 2 | 3
  Black, Not of Hispanic-American Origin | 1 | 1 | 2
  Hispanic-American | 0 | 0 | 0
  White, not of Hispanic-American Origin | 10 | 21 | 31
  Other or Unknown | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 14 | 22
  Germany | 5 | 8 | 13
  Italy | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders (Primary Medical Treatment in Arm 1, Primary Surgical Treatment in Arm 2)
Description: Nadir growth hormone <1 ng/mL during a standard 2 hour oral glucose tolerance test using 75 g glucose and normal IGF-I according to age and gender-matched standards.
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Treatment by Octreotide LAR | Surgical Debulking Followed by Octreotide LAR
Number analyzed (Participants) | 15 | 26
percentage of participants | 6.7 [.2 to 31.9] | 50 [29.9 to 70.1]

2. Primary Outcome: Percentage of Responders (All Treatments)
Description: as for outcome 1
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Treatment by Octreotide LAR | Surgical Debulking Followed by Octreotide LAR
Number analyzed (Participants) | 15 | 26
percentage of participants | 6.7 [.2 to 31.9] | 76.9 [56.4 to 91]

3. Secondary Outcome: Percentage of Responders (Only Including Surgical Failures in Arm 2)
Description: as for outcome 1
Time Frame: 3 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Medical Treatment by Octreotide LAR | Surgical Debulking Followed by Octreotide LAR
Number analyzed (Participants) | 15 | 13
percentage of participants | 6.7 [.2 to 31.9] | 53.9 [25.1 to 80.8]

ADVERSE EVENTS:
Arm/Group | Medical Treatment by Octreotide LAR | Surgical Debulking Followed by Octreotide LAR
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/26
Other Adverse Events (participants affected / at risk) | 5/15 | 12/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Treatment by Octreotide LAR (N=15) | Surgical Debulking Followed by Octreotide LAR (N=26)
Hyponatremia with Abdominal Discomfort (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Medical Treatment by Octreotide LAR (N=15) | Surgical Debulking Followed by Octreotide LAR (N=26)
Nausea/Vomiting/Diarrhea/Bloating/Constipation/GI distress (Gastrointestinal disorders) | 2 (7) | 9 (19)
Headaches (Nervous system disorders) | 1 (1) | 6 (7)
Pain at the Injection site (Surgical and medical procedures) | 0 (0) | 2 (2)
Otitis Media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Seizures (Seizure disorder since childhood) (Nervous system disorders) | 1 (1) | 0 (0)
Dry nose (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory Infections/Cold symptoms/ Cough (Infections and infestations) | 0 (0) | 2 (5)
Sinus irritation/pressure (General disorders) | 0 (0) | 2 (2)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 3 (3)
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Arm Weakness/Numbing (General disorders) | 0 (0) | 1 (2)
Muscle ache (General disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Planned excision of occipital skin tumor (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes